CLINICAL TRIAL: NCT06483932
Title: Effect of Dried Barberry Consumption on Cardiometabolic Risk Factors in Individuals With Mild to Moderate Hypertriglyceridemia
Brief Title: Barberry and Cardiometabolic Risk Factors in Individuals With Hypertriglyceridemia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Shahid Beheshti University (Other)
Collaborators: Shahid Beheshti University of Medical Sciences (Other); Kashan University of Medical Sciences (Other)
Responsible Party: Principal Investigator, Javad Nasrollahzadeh, Associate Professor, Shahid Beheshti University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 43008122
Record Dates: First submitted 2024-06-26; First posted 2024-07-03 (Actual); Last update posted 2025-05-06 (Actual); Status verified 2024-12

CONDITIONS: Hyperlipidemias; Hypertriglyceridemia
MeSH Terms: conditions — Hyperlipidemias; Hypertriglyceridemia | interventions — Caloric Restriction

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Control (Active Comparator): A diet with a reduced calorie intake
  Interventions: Other: Low-calorie diet
- Barberry (Experimental): A diet with a reduced calorie intake, coupled with the consumption of barberry
  Interventions: Other: Dried barberry; Other: Low-calorie diet

INTERVENTIONS:
Other: Dried barberry — Subjects will ingest 10 grams of powdered seedless barberry on a daily basis, in conjunction with the low-calorie diet.
  Other Names: Berberis vulgaris
  Arms: Barberry
Other: Low-calorie diet — Diet with 500 kcal subtracted from the daily energy requirement

SUMMARY:
Barberry is a well-documented medicinal plant that is utilized as a feed additive in a variety of food cultures. Barberry is a rich source of antioxidants, minerals, phenolic compounds, and flavonoids. Based on the results of animal and human studies, barberry may have therapeutic and medicinal properties, including the ability to improve blood lipid profile. The present study will investigate the effect of seedless barberry consumption on cardiometabolic factors in overweight or obese individuals with mild to moderate hypertriglyceridemia.

DETAILED DESCRIPTION:
This study is an open-label, randomized, controlled clinical trial and will recruit those who are willing to participate and meet the inclusion criteria. Inclusion criteria are fasting serum triglycerides 150-499 mg/dL, body mass index 25-40 kg/m2, age range 18-75 years. Exclusion criteria are regular use of drugs of the fibrate family, regular use of fish oil supplements or omega-3 supplements or flax seed or chia seed, treatment with glucocorticoids, end-stage renal disease. Subjects who agree to participate in the study will be randomly assigned to one of two study groups. All patients in both groups will be prescribed a low-calorie diet. In the first group, 10 grams of powdered seedless barberry will be consumed daily in addition to the low-calorie diet. The second group (control group) will continue with the low calorie diet. The study will last 8 weeks. Patients are asked to refrain from using over-the-counter herbal medicines and dietary supplements during the study. A baseline fasting blood sample, blood pressure measurements, and anthropometric indices will be obtained. Subsequent assessments will be made at four-week and eight-week intervals.

ELIGIBILITY:
Inclusion Criteria:

* Fasting serum triglycerides 150-499 mg/dL,
* Body mass index 25-40 kg/m2
* Age range 18-75 years

Exclusion Criteria:

* Regular use of drugs of the fibrate family, fish oil supplements or omega-3 supplements
* Regular consumption of flax seed or chia seed
* Treatment with glucocorticoids
* End-stage renal disease

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2024-09-09 (Actual); Primary Completion 2025-03-01 (Actual); Study Completion 2025-05-01 (Actual)

PRIMARY OUTCOMES:
Plasma concentration of triglycerides | At baseline, the fourth week and the eighth week of study
  The plasma triglyceride concentration 12 hours after the subjects had fasted
Plasma concentration of high-density lipoprotein cholesterol (HDL-C) | At baseline, the fourth week and the eighth week of study
  The plasma HDL-C concentration 12 hours after the subjects had fasted

SECONDARY OUTCOMES:
Body weight | At baseline, the fourth week and the eighth week of study
  Body wight loss (kg)
Plasma Cholesterol | At baseline, the fourth week and the eighth week of study
  The plasma total cholesterol and LDL-C concentrations 12 hours after the subjects had fasted
Plasma proprotein convertase subtilisin/kexin type 9 (PCSK9) | At baseline and the eighth week of study
  The plasma PCSK9 concentration 12 hours after the subjects had fasted
Plasma C-reactive protein | At baseline and the eighth week of study
  The plasma CRP concentration
Plasma Insulin | At baseline and the eighth week of study
  The plasma insulin concentration 12 hours after the subjects had fasted
Blood pressure | At baseline, the fourth week and the eighth week of study
  Systolic and diastolic bliood pressure
Urinary polyphenol | At baseline, the fourth week and the eighth week of study
  Total polyphenol concentration in spot urine sample

CONTACTS AND LOCATIONS:
Overall Officials: Javad Nasrollahzadeh, Ph.D, Principal Investigator — Shahid Beheshti University of Medical Sciences
Locations (1):
- Shahid Beheshty Unversity Hospital, Kāshān, Isfahan, Iran

IPD SHARING:
Plan to Share IPD: No